CLINICAL TRIAL: NCT03580668
Title: Multi-center, Canadian, Non-interventional, Cohort Study of the Effectiveness, Safety, Adherence, and Health-related Quality of Life in HIV-1 Infected Adult Patients Receiving Bictegravir/ Emtricitabine/Tenofovir Alafenamide (B/F/TAF)
Brief Title: Effectiveness, Safety, Adherence, and Health-related Quality of Life in HIV-1 Infected Adults Receiving Bictegravir/ Emtricitabine/Tenofovir Alafenamide
Acronym: BIC-STaR
Status: Completed | Type: Observational
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: GS-CA-380-4574
Record Dates: First submitted 2018-06-26; First posted 2018-07-09 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: HIV-1-infection
Keywords: Observational
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- B/F/TAF: Bictegravir/Emtricitabine/Tenofovir alafenamide (B/F/TAF) therapy in HIV-1 infected adults who initiate B/F/TAF therapy
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — B/F/TAF administered in accordance with the approved product monograph
  Other Names: Biktarvy®

SUMMARY:
The primary objective of this study is to evaluate HIV-1 RNA suppression, defined as HIV-1 RNA <50 copies/mL, at 12 months after initiating or switching to Bictegravir/ Emtricitabine/Tenofovir alafenamide (B/F/TAF).

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Signed informed consent
* Initiating treatment with B/F/TAF in accordance with the product monograph

Exclusion Criteria:

Participation in any other observational or interventional clinical trial without prior approval from the Medical Monitor

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of ART-naïve and ART-experienced HIV-1 infected adults aged ≥18 years initiating treatment with B/F/TAF in routine clinical care in Canada.
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 12 Months after initiating or switching to B/F/TAF | 12 months

SECONDARY OUTCOMES:
Proportion of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 3 Months after initiating or switching to B/F/TAF | 3 months
Proportion of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 6 Months after initiating or switching to B/F/TAF | 6 months
Proportion of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 24 Months after initiating or switching to B/F/TAF | 24 months
Proportion of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 36 Months after initiating or switching to B/F/TAF | 36 months
Proportion of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 48 Months after initiating or switching to B/F/TAF | 48 months
Proportion of Participants with HIV-1 RNA Suppression (HIV RNA < 50 copies/mL) at 60 Months after initiating or switching to B/F/TAF | 60 months
Change in CD4 Cell Count at 3 Months | 3 months
Change in CD4 Cell Count at 6 Months | 6 months
Change in CD4 Cell Count at 12 Months | 12 months
Change in CD4 Cell Count at 24 Months | 24 months
Change in CD4 Cell Count at 36 Months | 36 months
Change in CD4 Cell Count at 48 Months | 48 months
Change in CD4 Cell Count at 60 Months | 60 months
CD4/CD8 Ratio at 3 Months | 3 months
CD4/CD8 Ratio at 6 Months | 6 months
CD4/CD8 Ratio at 12 Months | 12 months
CD4/CD8 Ratio at 24 Months | 24 months
CD4/CD8 Ratio at 36 Months | 36 months
CD4/CD8 Ratio at 48 Months | 48 months
CD4/CD8 Ratio at 60 Months | 60 months
Proportion of Participants Experiencing Adverse Events (AEs) | 60 months
Proportion of Participants Experiencing and Serious Adverse Events (SAEs) | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- Canada (6):
  - Clinique Medicale du Quartier Latin, Montreal
  - University of Ottawa, Ottawa
  - Regina General Hospital, Regina
  - St. Clair Medical Association/Balmoral Clinic, Toronto
  - Maple Leaf Research, Toronto
  - Spectrum Health, Vancouver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Antinori A, Yokomaku Y, Elinav H, Pullukcu H, de Wet J, Antela A, Lu PL, Sabranski M, Kim YS, Bonnet F, den Hollander J, Jackson A, Choy CY, Cai W, Zhang F, Thorpe D, Marongiu A, Harrison R, Jarrett J, Boffito M. Quality of Life and Treatment Satisfaction in People with HIV Switching to Bictegravir/Emtricitabine/Tenofovir Alafenamide: Pooled Analysis from Observational Cohort Studies. Infect Dis Ther. 2026 Jan;15(1):217-244. doi: 10.1007/s40121-025-01252-w. Epub 2025 Nov 24. PMID 41284214
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-CA-380-4574